CLINICAL TRIAL: NCT03826459
Title: The PICS Trial: A Pilot Randomized Controlled Trial of Non-Locked vs. Locked Uterine Closure at Cesarean Section for Prevention of Uterine Isthmocele Formation
Brief Title: Preventing Isthmocele After Cesarean Section
Acronym: (PICS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Mara Sobel, Obstetrician/Gynecologist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PICS
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Cesarean Section Complications; Uterine Scar Diverticulum; Uterine Scar From Previous Cesarean Delivery

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either locked or non-locked uterine closure at the time of cesarean section.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locked Uterine Closure (Active Comparator): Participants will undergo two-layer closure of the hysterotomy site at the time of cesarean section. The first layer will use a running & locking technique. The second layer will be performed based on surgeon preference.
  Interventions: Procedure: Locked Uterine Closure
- Non-Locking Uterine Closure (Experimental): Participants will undergo two-layer closure of the hysterotomy site at the time of cesarean section. The first layer will use a running & non-locking technique. The second layer will be performed based on surgeon preference, but cannot be of a locking technique.
  Interventions: Procedure: Non-Locking Uterine Closure

INTERVENTIONS:
Procedure: Non-Locking Uterine Closure — The first layer of the two-layer uterine closure will be sutured with a running & non-locking technique. The second layer cannot be of a locking technique.
  Arms: Non-Locking Uterine Closure
Procedure: Locked Uterine Closure — The first layer of the two-layer uterine closure will be sutured with a running & locking technique. The second layer can be locking or non-locking.
  Arms: Locked Uterine Closure

SUMMARY:
Cesarean section accounts for nearly 30% of births in Canada, and is the most commonly performed surgery by Obstetrician Gynecologists. Cesarean scar isthmocele, meaning a defect in the uterine wall at the site of a previous uterine incision, is a common complication of this surgery. While most are likely asymptomatic, isthmoceles can lead to major complications in pregnancy (uterine rupture, invasive placentation, cesarean scar ectopic pregnancy) and outside of pregnancy (abnormal uterine bleeding, infertility and pain). Studies have shown that the method used to suture the uterus at the time of a cesarean section may have an impact on the incidence of post-operative isthmocele formation. Our study is a randomized control trial of the impact of locked vs unlocked uterine closure at cesarean section on the incidence of isthmocele formation. Women undergoing cesarean section will be randomized to have either a locked or unlocked uterine closure. They will then return 6 months after their surgery for a transvaginal ultrasound to evaluate the presence or absence of an isthmocele.

This study is a pilot trial. The investigators hope to determine the feasibility of completing a large randomized control trial by recording: a) the number of patient who agree to participate in this study, b) the number of patients who receive the correct intervention and, c) the number of patients who return for their post operative ultrasound.

The investigators also plan to assess multiple secondary outcomes. First, the goal is to determine the isthmocele incidence within the study subjects of the pilot trial in order to perform a power calculation for a subsequent larger trial in this area. Another goal is to determine if the uterine closure techniques in this study lead to differences in surgical time, blood loss or the need for intra- or post-operative blood transfusion. Last, the study will collect data on the suture material most commonly used in this study to determine if this requires standardization in the subsequent larger trial.

DETAILED DESCRIPTION:
Cesarean section accounts for nearly 30% of all deliveries in Canada, and is the most commonly performed surgery by Obstetrician Gynecologists (OBGYNs) in Canada. Therefore, it is important to understand the short and long-term complications of this procedure. Recently, emphasis has been placed on cesarean scar isthmocele as a long-term complication. An isthmocele is a defect at the cesarean section scar site with a depth of at least 1-2mm. Isthmoceles can lead to major obstetrical complications such as cesarean scar pregnancy, invasive placentation, and uterine rupture. More commonly, patients present with gynecologic symptoms: abnormal uterine bleeding, pain, and infertility. Up to 30-50% of patients with an isthmocele report symptoms when inquired. Isthmoceles have an incidence of 19-88% following cesarean section. This wide range is due to discrepancies in study technique, diagnostic criteria, and patient characteristics.

While medical and surgical treatment options are available for cesarean scar isthmocele, our focus should turn to prevention at the time of cesarean section. Evidence suggests double-layer (vs. single-layer) uterine closure decreases the formation of cesarean scar isthmocele and increases residual myometrial thickness (RMT). Additionally, uterine closure with a locked suturing technique may result in greater isthmocele depth and size, and a thinner RMT at the cesarean scar site. To our knowledge however, no study has determined the impact of a locked vs. unlocked double-layer closure technique on isthmocele prevention. Locked sutures, believed to be more hemostatic, may cause tissue necrosis and impair wound healing. Interestingly, evidence does not support reductions in operative blood loss with locked closure techniques. The hypothesis is that unlocked double-layer uterine closure can reduce isthmocele formation and thus improve longterm maternal outcomes without impacting operative blood loss or other short-term surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing their first cesarean section

Exclusion Criteria:

* previous uterine hysterotomy (caesarean section, myomectomy, etc.)
* known uterine anomalies
* active labour
* known bleeding disorder
* maternal connective tissue disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since this is a study done at the time of cesarean section, only females are eligible.
Enrollment: 41 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants Enrolled | 6 months
  Number of potential participants approached who actually enrolled in the trial
Number of Participants that Cross-Over | 6 months
  Number of participants who cross-over to the other study arm (i.e. who receive the incorrect uterine closure technique)
Number of Participants Lost to Follow Up | 6 months
  Number of participants enrolled in the trial who do not present for their follow up ultrasound at 6 months.

SECONDARY OUTCOMES:
Incidence of Isthmocele | 6 months
  The presence of an isthmocele (minimum 2 mm x 2 mm) identified on a transvaginal ultrasound 6 months after the cesarean section
Estimated Blood Loss | Through surgery completion (estimated 1 hour)
  Number of mL of blood lost at the time of cesarean section
Change in Hemoglobin | 24 hours
  Change in Hgb from pre-operative measurement to Hgb measurement on post-operative day #1
Operative Time | Through surgery completion (estimated 1 hour)
  Length of surgery (minutes)
Number of Blood Transfusions | Throughout hospital stay (estimated 48 hours)
  Number of intraoperative and post-operative blood transfusions given to each participant
Additional Hemostatic Sutures | Start to end of surgery
  Number of additional hemostatic sutures placed in the uterus for each participant
Suture Material | 6 months
  Type of suture material used for hysterotomy closure
Use of Additional Oxytocin in Units | Throughout hospital stay (estimated 48 hours)
  Number of units of additional oxytocin given to each participant as a uterotonic agent (beyond usual dose of intraoperative oxytocin)
Use of Ergotamine in mg | Throughout hospital stay (estimated 48 hours)
  Number of mg Ergotamine used as a uterotonic agent, if required
Use of Hemabate in mg | Throughout hospital stay (estimated 48 hours)
  Number of mg Ergotamine used as a uterotonic agent, if required
Use of Misoprostol in mcg | Throughout hospital stay (estimated 48 hours)
  Number of mcg Misoprostol used as a uterotonic agent, if required

CONTACTS AND LOCATIONS:
Overall Officials: Mara Sobel, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warshafsky C, Kirubarajan A, Chaikof M, Stere A, Chudawala U, Li Q, Huszti E, Mohamed D, Abdalla MH, Hartman A, Sanders A, Murji A, Sobel M. Preventing Isthmocele After Cesarean Section (PICS): A Pilot Randomized Controlled Trial. J Obstet Gynaecol Can. 2022 Nov;44(11):1134-1135. doi: 10.1016/j.jogc.2022.08.003. Epub 2022 Aug 12. No abstract available. PMID 35970439